CLINICAL TRIAL: NCT01728662
Title: Post Market Investigator Sponsored Study of Emphysematous Lung Sealant Therapy in Homogeneous Emphysema Using a Modified Treatment Strategy
Brief Title: Emphysematous Lung Sealant Therapy in Homogeneous Emphysema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC127000 CTIL
Record Dates: First submitted 2012-10-23; First posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Patients With Advanced Homogeneous Emphysema
Keywords: emphysema; lung volume reduction therapy
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ELVR Procedure (Experimental): A single subsegmental AeriSeal System treatment consists of the administration of 10 mL Foam Sealant administered through a standard fiberoptic bronchoscope via an administration syringe and bronchoscopic catheter into the target area of damaged lung
  Interventions: Procedure: ELVR Procedure

INTERVENTIONS:
Procedure: ELVR Procedure — Lung Volume Reduction Procedure

SUMMARY:
This study will test that hypothesis that endoscopic lung volume reduction therapy performed using emphysematous lung sealant treatment can be improved using smaller doses delivered to more a larger number of treatment sites.

DETAILED DESCRIPTION:
This is an investigational, single arm, physician-sponsored study that will be conducted at Rabin Medical Center under the direction of Professor Mordechai Kramer. Patients will receive AeriSeal System therapy using a new treatment algorithm to deliver approved foam sealant components at doses at or below those previously shown to be safe and effective during prior studies. Investigational aspects of this study involve only the method of administration of material, not the material itself. The specific modifications to the treatment method proposed in this study include: 1) lowering the dose per subsegment of AeriSeal System Foam Sealant to 10 mL from the approved 20 mL dose; 2) administering the subsegmental doses at more anatomic locations with the goal of improving distribution of material and achieving more effective lung volume reduction; 3) eliminating the administration of air through the instrument channel of the bronchoscope following Foam Sealant delivery to simply and shorten the procedure, improving safety.

The study is designed to treat 8 patients. The first 4 patients will receive treatment with 10 mL of AeriSeal System Foam Sealant administered at 6 subsegments, 3 in each upper lobe (a dose of 60 mL of AeriSeal Foam Sealant). This group will be followed until all 4 have completed 1 month (28 day) follow-up. A safety review of the data will then be conducted prior to initiating treatment in the next group of 4 patients. This review will include an assessment of adverse events and physiological responses.

Assuming no emergent safety issues are identified, the next group of 4 patients will receive treatment with 10 mL of AeriSeal System Foam Sealant administered at 8 subsegments, 3 in each upper lobe, one in the upper-most portion of the right middle lobe, one in the upper-most portion of the lingual (a dose of 80 mL of AeriSeal Foam Sealant).

All patients will be followed for 24 weeks after completion of therapy and receive standard medical treatment in addition to treatment with the AeriSeal System.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of GOLD Stage III/IV homogeneous emphysema
2. FEV1/FVC <70 % predicted, FEV1 of < 50% predicted, TLC > 100% of predicted, and RV > 150% predicted.
3. chest CT scan showing evidence of tissue destruction indicative of homogeneous (uniformly distributed) emphysema.
4. Patients must also have ≤ 15% perfusion in both upper lobes on a quantitative lung perfusion scan indicating bilateral target sites for therapy.
5. Patients must be > 40 years of age.

Exclusion Criteria:

1. Alpha-1 antitrypsin deficient patients (i.e. those with serum levels < 80 mg/dL, or < 11 µmol/L or 57 mg/dL).
2. patients who are pregnant or breast feeding.
3. patients who are smoking.
4. patients using other investigational medications will be excluded.
5. Patients must have persistent symptoms despite medical therapy and either not be candidates for Lung Volume Reduction Surgery (LVRS) or have elected not to undergo LVRS.
6. have no significant co-morbid conditions that could influence study outcomes or their ability to tolerate bronchoscopy.
7. Specifically, patients should not have a history of prior major thoracic surgery, HIV infection, clinically significant asthma, bronchiectasis, pulmonary hypertension or coronary heart disease.
8. Patients must also not be dependent on medications that could increase the risk of undergoing treatment or adversely effect the chance of recovering from treatment (i.e. high dose steroids, immunosuppressive agents, or anticoagulants)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Overall safety assessment | 6 months
  Overall assessment of safety based on review
  1. Clinical and laboratory results:
     * Serious Adverse Events (SAEs)
     * Serious Adverse Device Effects (SADEs)
     * Unanticipated Serious Adverse Device Effects (USADEs)
     * Physical Examinations
     * Vital signs
     * Serum chemistry and hematology.
  2. Changes from baseline in clinical pathology or lung physiology based on:
     * Blood gases
     * Pulmonary function data
     * Radiology data

SECONDARY OUTCOMES:
Efficacy Evaluations will include: | 6 months
  * CT evidence of lobar volume reduction at site(s) of AeriSeal administration at 12 weeks assessed quantitatively by digital integration of CT dicom images collected using a standardized image acquisition and reconstruction algorithm.
  * Change from baseline at 12 and 24 weeks in RV/TLC
  * Change from baseline at 12 and 24 weeks in FEV1
  * Change from baseline at 12 and 24 weeks in FVC
  * Change from baseline at 12 and 24 weeks in 6 MWT
  * Change from baseline at 12 and 24 weeks in MRCD score
  * Change from baseline at 12 and 24 weeks in SGRQ total domain score

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai R Kramer, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel